CLINICAL TRIAL: NCT00232024
Title: Assessment of Efficacy and Safety of Tegaserod Treatment and Placebo in Women With Dyspepsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919D2301
Record Dates: First submitted 2005-09-08; First posted 2005-10-04 (Estimated); Last update posted 2008-02-01 (Estimated); Status verified 2008-01

CONDITIONS: Dyspepsia
Keywords: Dyspepsia, gastrointestinal, tegaserod
MeSH Terms: conditions — Dyspepsia | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
This study is being done to evaluate the safety, tolerability and satisfactory relief of dyspepsia symptoms in females excluding those with predominant stomach pain. Tegaserod will be evaluated at 6mg twice daily and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 years or older
* Self-reported presence of persistent or recurrent adverse digestive symptoms consistent with dyspepsia for at least 12 weeks, not necessarily consecutive, during the previous 12 months.

Exclusion Criteria:

* Abnormal upper GI endoscopy findings such as esophageal, gastric erosions or ulcers and/or duodenal ulcers/erosions.
* Any of the following symptoms: heartburn, epigastric pain, nausea or vomiting.

Other protocol-defined inclusion/exclusion criteria may appl

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 1296
Dates: Start 2004-01; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Over 6 weeks of treatment assessment of percent of days with satisfactory relief of dyspepsia and/or average severity score in (average of post-prandial fullness early satiety and bloating)

SECONDARY OUTCOMES:
Average severity score during each week.
Percentage of days with satisfactory relief of dyspepsia during each week.
Weekly global assessment of change in dyspepsia condition.
Daily assessment of improvment of individual symptoms postprandial fullness early satiety, bloating, abdominal pain, nausea and vomiting.
Quality of life at end of treatment compared to baseline.
Safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Basel
Locations (1):
- Novartis, East Hanover, New Jersey, United States